CLINICAL TRIAL: NCT02341599
Title: A Phase 1, Non-randomized, Parallel-group, Open-label Study to Characterize the Pharmacokinetics of a Single Intravenous Dose of CB-238,618 in Subjects With Varying Degrees of Renal Impairment Compared to Healthy Subjects
Brief Title: Study of Pharmacokinetics of a Single IV Dose of CB-238,618 in Subjects With Varying Degrees of Renal Impairment Compared to Healthy Subjects (MK-6183-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6183-001; 618-REN-14-02 (Other: Cubist Study Number); MK-6183-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-12-12; First posted 2015-01-19 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A: Healthy (Experimental): Healthy participants with normal renal function (Stage 1: eGFR ≥90 mL/min/1.73m^2).
  Interventions: Drug: MK-6183
- Group B: Mild RI (Experimental): Participants with mild RI (Stage 2: eGFR ≥60 to <90 mL/min/1.73m^2).
  Interventions: Drug: MK-6183
- Group C: Moderate RI (Experimental): Participants with moderate RI (Stage 3: eGFR ≥30 to <60 mL/min/1.73m^2).
  Interventions: Drug: MK-6183
- Group D: Severe RI (Experimental): Participants with severe RI (Stage 4: eGFR <30 mL/min/1.73m^2) not receiving HD.
  Interventions: Drug: MK-6183
- Group E: ESRD-HD (Experimental): Participants with ESRD who are receiving HD for at least 3 months preceding the initial dose in this study (Stage 5).
  Interventions: Drug: MK-6183

INTERVENTIONS:
Drug: MK-6183 — MK-6183 (CB-238,614) is supplied as lyophilized powder 500 mg vial and mixed into solution for 100 mL intravenous (IV) administration over 1 hour.
  Other Names: CB-238,618

SUMMARY:
The purpose of this study is to characterize the effect of renal function on the plasma, urine, and dialysate pharmacokinetic profile of MK-6183 (CB-238,618) in humans. The study will also assess the safety profile and tolerability of MK-6183 in healthy participants, participants with varying degrees of renal impairment (RI), or participants with end-stage renal disease (ESRD) requiring hemodialysis (HD), based on estimated glomerular filtration rate (eGFR).

ELIGIBILITY:
Inclusion Criteria:

* Participants who are healthy; or who have mild, moderate, or severe RI; or who have ESRD requiring HD. Participants with ESRD requiring HD should have been receiving HD 3 times per week for at least 3 months preceding the initial dose in this study

Exclusion Criteria:

* For healthy participants (Group A): history or presence of any clinically significant illness (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, musculoskeletal, or psychiatric) or any other condition, including clinically significant anemia, which in the opinion of the investigator would jeopardize the safety of the participant or the validity of the study results
* For participants with RI (Groups B to E): as above, except that RI and other medical conditions commonly associated with renal impairment (eg, hypertension, diabetes, which should be stable for at least three months preceding the initial dose of study medication in this study) are allowed
* Clinically significant abnormalities on physical examination, medical history, 12-lead electrocardiogram (ECG), vital signs, or laboratory values, as judged by the investigator or designee. Subjects with renal impairment should have clinical laboratory values consistent with their disease and approved by the investigator
* Evidence of clinically significant hepatic impairment including alanine aminotransferase or aspartate aminotransferase >1.5 × upper limit of normal (ULN) or bilirubin >1 × ULN
* Hemoglobin <8 g/dL, unless considered stable and not clinically significant in the opinion of the investigator in subjects with ESRD and on HD
* Participants with renal impairment who are not on a chronic stable drug regimen, defined as starting a new drug or changing dosage within 14 days prior to administration of study medication, except for drugs administered in relationship to HD
* Participants with fluctuating or rapidly deteriorating renal function (assessment of the stability of the subject's renal function will be determined by the investigator)
* Participant has a currently functioning renal transplant and/or has been on significant immunosuppressant therapy, as determined by the investigator, within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2015-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants, participants with varying degrees of renal impairment (RI), and participants with end-stage renal disease (ESRD) requiring hemodialysis (HD) (renal status was based on estimated glomerular filtration rate [eGFR]) were recruited at 2 study sites in the United States.
Groups:
- Group A: Healthy: Healthy participants with normal renal function (Stage 1: eGFR ≥90 mL/min/1.73m^2) received MK-6183 1 g as a 1-hour IV infusion.
- Group B: Mild RI: Participants with mild RI (Stage 2: eGFR ≥60 to <90 mL/min/1.73m^2) received MK-6183 1 g as a 1-hour IV infusion.
- Group C: Moderate RI: Participants with moderate RI (Stage 3: eGFR ≥30 to <60 mL/min/1.73m^2) received MK-6183 500 mg as a 1-hour IV infusion.
- Group D: Severe RI: Participants with severe RI (Stage 4: eGFR <30 mL/min/1.73m^2 [not receiving HD]) received MK-6183 500 mg as a 1-hour IV infusion.
- Group E: ESRD-HD: Participants with ESRD who underwent HD for at least 3 months preceding the initial dose in this study (Stage 5) received MK-6183 250 mg as a 1-hour infusion twice (once prior to HD and once after HD [doses given 48 hours apart]).
Period: Overall Study
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD
Started | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (2.43) | 63.8 (11.16) | 69.1 (4.88) | 65.3 (10.47) | 55.1 (7.55) | 61.7 (44.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 4 | 1 | 11
  Male | 6 | 5 | 7 | 4 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Dosing to Last Measurable Concentration (AUC0-last) of MK-6183
Description: AUC0-last is the area under the plasma concentration-time curve from the time of dosing to the last post-dose measurable concentration. Blood samples for Group E were collected both prior to and during HD (Period 1) and after HD (Period 2) [data from Periods 1 and 2 were analyzed separately]. In Period 1, HD commenced 3.5 hours post-dose (HD duration was 3.5 to 4 hours) and sample collection continued until 48 hours post-dose. The specific time frame of plasma sample collection for Group E: Period 1 was pre-dose, 0.5 hours post-dose, EOI, 1.5 hours post-dose, 2 hours post-dose, 3 hours post-dose (pre-HD), 3.5 hours post-dose with HD, 5 hours post-dose with HD, pre-end of HD, 30 min post-HD, 1 hour post-HD, 2 hours post-HD, 12 hours post-dose, 24 hours post-dose, and 48 hours post-dose.
Time Frame: Groups A to D & Group E: Period 2: Pre-dose and 0.5, 1 (end of infusion; EOI), 1.5, 2, 3, 6, 12, 24, 48, and 72 hours post-dose
Population: All participants who received MK-6183 and had viable results are included. One participant from Group E: Period 1 and 1 participant from Group E: Period 2 were excluded due to implausible concentration values.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Groups:
- Group E: ESRD-HD Period 1: Participants with ESRD who underwent HD for at least 3 months preceding the initial dose of study drug (Stage 5) received CB-238,615 250 mg as a 1-hour infusion prior to undergoing HD in Period 1. Both plasma and dialysate samples were collected during Period 1.
- Group E: ESRD-HD Period 2: Participants with ESRD who underwent HD for at least 3 months preceding the initial dose of study drug (Stage 5) received CB,238-615 250 mg as a 1-hour infusion within 2 hours of completing HD in Period 2 (Period 2 HD commenced 2 days after completing Period 1 HD).
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1 | Group E: ESRD-HD Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 7
ug*hr/mL | 87.6 (8.49) | 114.8 (23.20) | 97.5 (25.71) | 228.0 (63.24) | 77.4 (8.79) | 270.6 (76.70)

2. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 12 days
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- Group E: ESRD-HD Periods 1 and 2: Participants with ESRD who underwent HD for at least 3 months preceding the initial dose of study drug (Stage 5) received CB-238,615 250 mg as 2 1-hour infusions (1 before HD and 1 after HD).
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Periods 1 and 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants | 4 | 2 | 2 | 3 | 4

3. Primary Outcome: AUC From Dosing to ∞ (AUC0-∞) of MK-6183
Description: AUC0-∞ is the extrapolated area under the plasma concentration-time curve from the time of dosing to infinity. Blood samples for Group E were collected both prior to and during HD (Period 1) and after HD (Period 2) [data from Periods 1 and 2 were analyzed separately]. In Period 1, HD commenced 3.5 hours post-dose (HD duration was 3.5 to 4 hours) and sample collection continued until 48 hours post-dose. The specific time frame of plasma sample collection for Group E: Period 1 was pre-dose, 0.5 hours post-dose, EOI, 1.5 hours post-dose, 2 hours post-dose, 3 hours post-dose (pre-HD), 3.5 hours post-dose with HD, 5 hours post-dose with HD, pre-end of HD, 30 min post-HD, 1 hour post-HD, 2 hours post-HD, 12 hours post-dose, 24 hours post-dose, and 48 hours post-dose. For statistical analyses, Group A is the reference and least squares (LS) mean ratios for tests (Groups B to E) are calculated as test/reference; Group E: Period 1 and Group E: Period 2 were also compared.
Time Frame: Groups A to D & Group E: Period 2: Pre-dose and 0.5, EOI, 1.5, 2, 3, 6, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1 | Group E: ESRD-HD Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 7
ug*hr/mL | 87.8 (8.43) | 115.1 (23.44) | 97.8 (25.70) | 228.6 (63.44) | 86.8 (7.63) | 296.3 (78.66)
Statistical Analysis 1: Comparison: Group A: Healthy vs Group B: Mild RI; Test type: Other — LS mean ratio of Group B/Group A; LS mean ratio = 1.29, 90% CI 2-sided [1.06 to 1.58] — LS mean ratio was calculated from analysis of variance (ANOVA) model
Statistical Analysis 2: Comparison: Group A: Healthy vs Group C: Moderate RI; Test type: Other — LS mean ratio of Group C/Group A; LS mean ratio = 1.08, 90% CI 2-sided [0.889 to 1.32] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 3: Comparison: Group A: Healthy vs Group D: Severe RI; Test type: Other — LS mean ratio of Group D/Group A; LS mean ratio = 2.51, 90% CI 2-sided [2.06 to 3.06] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 4: Comparison: Group A: Healthy vs Group E: ESRD-HD Period 1; Test type: Other — LS mean ratio of Group E: Period 1/Group A; LS mean ratio = 0.989, 90% CI 2-sided [0.806 to 1.21] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 5: Comparison: Group A: Healthy vs Group E: ESRD-HD Period 2; Test type: Other — LS mean ratio of Group E: Period 2/Group A; LS mean ratio = 3.27, 90% CI 2-sided [2.67 to 4.02] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 6: Comparison: Group E: ESRD-HD Period 1 vs Group E: ESRD-HD Period 2; Test type: Other — LS mean ratio of Group E: Period 1/Group E: Period 2; LS mean ratio = 0.299, 90% CI 2-sided [0.236 to 0.378] — LS mean ratio was calculated from ANOVA model

4. Primary Outcome: Maximum Plasma Drug Concentration (Cmax) of MK-6183
Description: Cmax is the maximum observed post-dose drug concentration in plasma. Blood samples for Group E were collected both prior to and during HD (Period 1) and after HD (Period 2) [data from Periods 1 and 2 were analyzed separately]. In Period 1, HD commenced 3.5 hours post-dose (HD duration was 3.5 to 4 hours) and sample collection continued until 48 hours post-dose. The specific time frame of sample collection for Group E: Period 1 was pre-dose, 0.5 hours post-dose, EOI, 1.5 hours post-dose, 2 hours post-dose, 3 hours post-dose (pre-HD), 3.5 hours post-dose with HD, 5 hours post-dose with HD, pre-end of HD, 30 min post-HD, 1 hour post-HD, 2 hours post-HD, 12 hours post-dose, 24 hours post-dose, and 48 hours post-dose. For statistical analyses, Group A is the reference and LS mean ratios for tests (Groups B to E) are calculated as test/reference; Group E: Period 1 and Group E: Period 2 were also compared.
Time Frame: Groups A to D & Group E: Period 2: Pre-dose and 0.5, EOI, 1.5, 2, 3, 6, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1 | Group E: ESRD-HD Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 7
ug/mL | 45.3 (5.23) | 47.2 (8.19) | 24.2 (5.95) | 30.8 (3.90) | 12.9 (4.60) | 15.6 (6.59)
Statistical Analysis 1: Comparison: Group A: Healthy vs Group B: Mild RI; Test type: Other — LS mean ratio of Group B/Group A; LS mean ratio = 1.04, 90% CI 2-sided [0.846 to 1.27] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 2: Comparison: Group A: Healthy vs Group C: Moderate RI; Test type: Other — LS mean ratio of Group C/Group A; LS mean ratio = 0.524, 90% CI 2-sided [0.428 to 0.641] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 3: Comparison: Group A: Healthy vs Group D: Severe RI; Test type: Other — LS mean ratio of Group D/Group A; LS mean ratio = 0.678, 90% CI 2-sided [0.554 to 0.831] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 4: Comparison: Group A: Healthy vs Group E: ESRD-HD Period 1; Test type: Other — LS mean ratio of Group E: Period 1/Group A; LS mean ratio = 0.273, 90% CI 2-sided [0.221 to 0.336] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 5: Comparison: Group A: Healthy vs Group E: ESRD-HD Period 2; Test type: Other — LS mean ratio of Group E: Period 2/Group A; LS mean ratio = 0.326, 90% CI 2-sided [0.265 to 0.402] — LS mean ratio was calculated from ANOVA model
Statistical Analysis 6: Comparison: Group E: ESRD-HD Period 1 vs Group E: ESRD-HD Period 2; Test type: Other — LS mean ratio of Group E: Period 2/Group E: Period 1; LS mean ratio = 0.808, 90% CI 2-sided [0.650 to 1.00] — LS mean ratio was calculated from ANOVA model

5. Primary Outcome: Apparent Total Body Clearance of MK-6183 From Plasma (CL)
Description: CL is a measure of the clearance of drug from plasma via metabolism and excretion. Blood samples for Group E were collected both prior to and during HD (Period 1) and after HD (Period 2) [data from Periods 1 and 2 were analyzed separately]. In Period 1, HD commenced 3.5 hours post-dose (HD duration was 3.5 to 4 hours) and sample collection continued until 48 hours post-dose. The specific time frame of plasma sample collection for Group E: Period 1 was pre-dose, 0.5 hours post-dose, EOI, 1.5 hours post-dose, 2 hours post-dose, 3 hours post-dose (pre-HD), 3.5 hours post-dose with HD, 5 hours post-dose with HD, pre-end of HD, 30 min post-HD, 1 hour post-HD, 2 hours post-HD, 12 hours post-dose, 24 hours post-dose, and 48 hours post-dose.
Time Frame: Groups A to D & Group E: Period 2: Pre-dose and 0.5, EOI, 1.5, 2, 3, 6, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1 | Group E: ESRD-HD Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 7
L/hour | 11.5 (1.23) | 9.0 (1.65) | 5.5 (1.64) | 2.4 (0.96) | 2.9 (0.26) | 0.9 (0.30)

6. Primary Outcome: Volume of Distribution at Steady State (Vss) of MK-6183
Description: Vss is the apparent volume of distribution at steady state for MK-6183. Blood samples for Group E were collected both prior to and during HD (Period 1) and after HD (Period 2) [data from Periods 1 and 2 were analyzed separately]. In Period 1, HD commenced 3.5 hours post-dose (HD duration was 3.5 to 4 hours) and sample collection continued until 48 hours post-dose. The specific time frame of sample collection for Group E: Period 1 was pre-dose, 0.5 hours post-dose, EOI, 1.5 hours post-dose, 2 hours post-dose, 3 hours post-dose (pre-HD), 3.5 hours post-dose with HD, 5 hours post-dose with HD, pre-end of HD, 30 min post-HD, 1 hour post-HD, 2 hours post-HD, 12 hours post-dose, 24 hours post-dose, and 48 hours post-dose.
Time Frame: Groups A to D & Group E: Period 2: Pre-dose and 0.5, EOI, 1.5, 2, 3, 6, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1 | Group E: ESRD-HD Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 7
Liters | 21.4 (2.64) | 22.8 (4.43) | 23.9 (6.03) | 19.4 (2.55) | 52.1 (16.57) | 25.3 (8.33)

7. Primary Outcome: Apparent Plasma Half-life (t½) of MK-6183
Description: t½ is the amount of time required for the plasma concentration of MK-6183 to reduce by 50%. Blood samples for Group E were collected both prior to and during HD (Period 1) and after HD (Period 2) [data from Periods 1 and 2 were analyzed separately]. In Period 1, HD commenced 3.5 hours post-dose (HD duration was 3.5 to 4 hours) and sample collection continued until 48 hours post-dose. The specific time frame of sample collection for Group E: Period 1 was pre-dose, 0.5 hours post-dose, EOI, 1.5 hours post-dose, 2 hours post-dose, 3 hours post-dose (pre-HD), 3.5 hours post-dose with HD, 5 hours post-dose with HD, pre-end of HD, 30 min post-HD, 1 hour post-HD, 2 hours post-HD, 12 hours post-dose, 24 hours post-dose, and 48 hours post-dose.
Time Frame: Groups A to D & Group E: Period 2: Pre-dose and 0.5, EOI, 1.5, 2, 3, 6, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1 | Group E: ESRD-HD Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 7
Hours | 2.1 (0.45) | 2.8 (0.33) | 4.0 (1.28) | 6.8 (1.90) | 18.1 (3.79) | 19.2 (5.04)

8. Secondary Outcome: Number of Participants Discontinuing From the Study Due to an AE
Description: as for outcome 2
Time Frame: Up to 12 days
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Periods 1 and 2
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Cumulative Amount of MK-6183 Excreted in Urine or Dialysate (Ae)
Description: Ae is the cumulative amount of drug excreted unchanged in urine or dialysate. For Groups A, B, C, and D, Ae was assessed in urine. For Group E: Period 1, Ae was assessed in dialysate (participants in Group E had no detectable urine data) at hourly collection intervals during HD (HD commenced 3 hours after dosing).
Time Frame: Groups A to D (urine): 0 to 24, 24 to 48, and 48 to 72 hours post-dose; Group E (dialysate): 0 to 1, 1 to 2, 2 to 3, and 3 to 4 hours after starting HD
Population: All participants who received MK-6183 and had viable results are included. For Group E, only results from Period 1 are presented as Period 2 sampling occurred post-HD.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1
Number analyzed (Participants) | 8 | 8 | 8 | 5 | 8
mg | 840.5 (65.33) | 699.1 (234.69) | 360.0 (33.82) | 309.1 (51.30) | 122.9 (29.21)

10. Primary Outcome: Renal Clearance of MK-6183 (CLr)
Description: CLr is the clearance of drug from plasma via the kidneys. Only data from Groups A, B, C, and D is presented; participants in Group E (Period 1) had no detectable urine data. Data for Group E: Period 1 are presented below in the dialysate clearance measure.
Time Frame: 0 to 24, 24 to 48, and 48 to 72 hours post-dose
Population: All participants who received MK-6183 and had viable results are included. CLr data are not presented for Group E.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI
Number analyzed (Participants) | 8 | 8 | 8 | 5
Liters/hour | 9.6 (1.14) | 6.1 (2.13) | 4.0 (1.61) | 1.7 (1.07)

11. Primary Outcome: Dialysate Clearance of MK-6183 (CLd)
Description: CLd is the amount of drug cleared from plasma via dialysis. Only data collected during HD (Group E: Period 1) is presented (HD commenced 3 hours after dosing).
Time Frame: 0 to 1, 1 to 2, 2 to 3, and 3 to 4 hours after starting HD
Population: All participants who received MK-6183 and had viable results are included. Only data for Group E: Period 1 is presented.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Group E: ESRD-HD Period 1
Number analyzed (Participants) | 8
Liters/hour | 1.4 (0.42)

12. Primary Outcome: Fraction of the Administered Dose of MK-6183 Excreted Unchanged in Urine or Dialysate (Fe)
Description: Fe is the fraction (percentage) of the administered dose that was excreted unchanged in urine (Groups A to D) or dialysate (Group E: Period 1; HD commenced 3 hours after dosing).
Time Frame: as for outcome 9
Population: All participants who received MK-6183 and had viable results are included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD Period 1
Number analyzed (Participants) | 8 | 8 | 8 | 5 | 8
mg | 84.0 (6.53) | 69.9 (23.47) | 72.0 (6.76) | 61.8 (10.26) | 49.2 (11.68)

ADVERSE EVENTS:
Time Frame: Up to 12 days
Description: All treated participants are included. Data from Group E: Period 1 and Group E: Period 2 are combined.
Arm/Group | Group A: Healthy | Group B: Mild RI | Group C: Moderate RI | Group D: Severe RI | Group E: ESRD-HD
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 2/8 | 2/8 | 3/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Healthy (N=8) | Group B: Mild RI (N=8) | Group C: Moderate RI (N=8) | Group D: Severe RI (N=8) | Group E: ESRD-HD (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnambulism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No